CLINICAL TRIAL: NCT02314858
Title: Tailored Treatment to Enhance Risk Perception in Sleep Apnea.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2809; R01HL120693 (NIH)
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Therapeutics; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Brief Personalized Video (BPV) (Experimental): Our BPV intervention focuses on augmenting risk perception and reducing optimistic bias by showing the patient a dramatic video of his/her own apnea (which shows them struggle to breathe), as well as by explaining the physiological processes involved in an apneic event. Specific apneic events are highlighted and associated decreases in blood oxygen levels are demonstrated via oxygen saturation recording superimposed on the video. This group will receive educational information about OSA, its consequences and the need for treatment.
  Interventions: Behavioral: Brief Personalized Video (BPV)
- Non-Personalized Video (NPV) (Active Comparator): NPV will include a video of someone having apnea, but it will not be personalized. This group will receive educational information about OSA, its consequences and the need for treatment.
  Interventions: Behavioral: Non-Personalized Video (NPV)
- Treatment As Usual (TAU) (Placebo Comparator): The TAU group will receive no special treatment from study interventionist team and will not view a video.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Brief Personalized Video (BPV) — The BPV group will view a portion of their own sleep study that took place during their overnight sleep study.
  Other Names: BPV
  Arms: Brief Personalized Video (BPV)
Behavioral: Non-Personalized Video (NPV) — The NPV group will see a stock video of someone with OSA.
  Other Names: NPV
  Arms: Non-Personalized Video (NPV)
Behavioral: Treatment as Usual (TAU) — The TAU group will not watch a video.
  Other Names: Standard of Care
  Arms: Treatment As Usual (TAU)

SUMMARY:
Obstructive Sleep Apnea (OSA) is seen in approximately 6% of Americans. It is a serious medical condition with significant medical and psychological consequences, including diabetes, hypertension, and cardiovascular disease. The treatment of choice for OSA is Positive Airway Pressure therapy (PAP). PAP supplies positive pressure to the upper airway creating a "pneumatic splint" to keep the airway open during sleep. Adherence to PAP is notoriously low, with as few as 50% reaching minimal guidelines for adherence. One comprehensive review of adherence research found that adherence to PAP was less than that for any other medical disorder. The problem of adherence is significant not only because of the medical consequences that can ensue, but also because third party payers have begun to refuse to pay for PAP therapy when adherence is less than optimal, even in the face of clinical improvement. This is a critical time to address this problem.

This research study is designed to identify methods that may help people respond to PAP, the most common therapy for OSA. Identifying these methods may be an important way to better care for patients with obstructive sleep apnea. With this research, the investigators hope to find ways to help people have a better response to treatment and a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Polysomnography (PSG) confirmed diagnosis of Obstructive Sleep Apnea (OSA)
* choice of PAP as preferred treatment
* judged by sleep physicians to be responders to PAP
* participants will be considered responders to PAP if they have an AHI of less than 5, do not snore, and have an arousal index of less than 10 when titrated to the proper pressure of PAP

Exclusion Criteria:

* Apnea-Hypopnea Index (AHI) < 15 on the diagnostic PSG and no daytime functional symptoms or associated cardiovascular disease
* a sleep disorder other than OSA that causes arousals from sleep (e.g., periodic limb movements, restless legs syndrome, insomnia)
* a current substance abuse problem
* a serious sleep-disruptive medical condition (e.g., end stage renal failure, severe Chronic Obstructive Pulmonary Disease (COPD), severe asthma)
* significant global cognitive impairment
* history of or current diagnosis of psychosis, bipolar disorder, or borderline, schizotypal or antisocial personality disorder, and uncontrolled depression or suicidal ideation
* change in antidepressant medications over the past 3 months
* women pregnant women, breast feeding, or planning on becoming pregnant
* currently enrolled in another research study

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Treatment Adherence | 90 days
  Treatment adherence as measured directly from the participant's PAP device. Adherence is monitored objectively as time at prescribed pressure and daily measures of adherence are transmitted remotely to the study site nightly using a wireless modem. There are several specific adherence measures that will be available from the PAP units. These include the average hours of use per night across all nights, the average hours of use on nights PAP is actually used, and the percentage of nights PAP is used across all nights.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Aloia, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States